CLINICAL TRIAL: NCT04007159
Title: A Human Repeat Insult Patch Test (HRIPT) in Healthy Subjects to Assess the Cutaneous Irritation and Sensitization Potential of Three Developmental Cosmetic Facial Products
Brief Title: To Evaluate Skin Irritation and Skin Sensitisation of Developmental Cosmetic Facial Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 212383
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Skin Care
Keywords: Skin Care, Cosmetic Facial Product
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The human repeated insult patch test (HRIPT) is a long standing, standard method to determine whether exposure to a topical product will elicit a cutaneous (dermal) irritant or allergic response (sensitization) under exaggerated (occluded) conditions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Developmental Serum (Experimental): The participants will be applied a semi-occlusive adhesive patch containing the developmental serum (0.02 milliliters per centimeters square [mL/cm^2] in an individual cell of the patch) topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 hours in weekdays and 72 hours in weekends) and for 48 hours (single application) in the challenge phase.
  Interventions: Other: Serum
- Developmental Lotion (Experimental): The participants will be applied a semi-occlusive adhesive patch containing the developmental lotion (0.02 mL/cm^2 in an individual cell of the patch) topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 hours in weekdays and 72 hours in weekends) and for 48 hours (single application) in the challenge phase.
  Interventions: Other: Lotion
- Developmental Cream (Experimental): The participants will be applied a semi-occlusive adhesive patch containing the developmental cream (0.02 mL/cm^2 in an individual cell of the patch) topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 hours in weekdays and 72 hours in weekends) and for 48 hours (single application) in the challenge phase.
  Interventions: Other: Cream
- Negative Control (Placebo Comparator): The participants will be applied a semi-occlusive adhesive patch containing the 0.9 percent (%) normal saline (0.02 mL/cm^2 in an individual cell of the patch) topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 hours in weekdays and 72 hours in weekends) and for 48 hours (single application) in the challenge phase.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Serum — Participants will be topically applied serum to the dorsum, under a semi-occlusive patch (0.02 milliliters per centimeters square [mL/cm^2] of serum in an individual cell of patch)
  Arms: Developmental Serum
Other: Lotion — Participants will be topically applied lotion to the dorsum, under a semi-occlusive patch (0.02mL/cm^2 of lotion in an individual cell of patch)
  Arms: Developmental Lotion
Other: Cream — Participants will be topically applied cream to the dorsum, under a semi-occlusive patch (0.02mL/cm^2 of cream in an individual cell of patch)
  Arms: Developmental Cream
Other: Normal Saline — Participants will be topically applied normal saline to the dorsum, under a semi-occlusive patch (0.02mL/cm^2 of normal saline in an individual cell of patch)
  Arms: Negative Control

SUMMARY:
The aim of this study is to assess irritant or allergic response of 3 developmental cosmetic facial products following a conventional human repeated insult patch test methodology for 6 weeks.

DETAILED DESCRIPTION:
A randomized, single blind (evaluator), single-center, Human Repeat Insult Patch Test (HRIPT) study in healthy adult participants aged 18 to 65 years to evaluate the cutaneous irritation and contact sensitization potential of 3 cosmetic facial skincare products. The participants will undergo repeated cutaneous application of semi-occlusive patch of 3 cosmetic facial skincare products and a reference product as a negative control (saline solution). HRIPT is a long standing, standard method to determine whether exposure to a topical product will elicit a cutaneous (dermal) irritant or allergic response (sensitization) under exaggerated (occluded) conditions. Screening of the participants will be performed at Visit 1 (i.e. from Day 0 to Day 14). The study will progress in 3-phases: Induction phase, Rest Phase and Challenge Phase. The Induction phase will continue for 3 consecutive weeks (Visit 2 to Visit 10); at visit 2, the area for patch application will be designated between the scapula and waistline, away from the spinal mid-line. A controlled amount (0.02 milliliters per centimeters square [mL/cm^2]) of each study product will be randomly assigned within the patch system of each participant into the appropriate separate cell (3 cells for each of the test products and 1 cell for the saline solution). Each patch will remain in place for 48 (± 4) hours on weekdays and 72 (± 4) hours on weekend. Induction phase will be followed by 2-week (Visit 11) Rest phase; where there will be no product or patch applications. Rest phase is further followed by Challenge phase at week 6 (Visit 12 to Visit 15) in which a naïve area of the skin will be selected and a new patch with each of the cells filled with study products will be applied. After 48 (±4) hours of patch application, participants will return to the site, the patch will be removed, and subsequent test-site evaluations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated in-formed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, with no clinically significant or relevant abnormalities in medical history or upon dermal examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant with Fitzpatrick phototype I to IV.
* A participant with healthy, intact skin at the proposed test area dorsum (below the shoulder, above the waist), as evaluated by a dermatologist, to ensure participant is free of clinically relevant dermatological conditions.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies involving investigational product(s) within 30 Days prior to study entry and/or during study participation.
* A participant who has participated in other studies including non-medicinal, cosmetic studies within 7 Days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant or intends to be-come pregnant during the study duration (self-reported).
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials/product (or closely related com-pounds) or any of their stated ingredients, to hypoallergenic tape, or to the cotton patches.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the Lifestyle Considerations; a) applying other product to test site, using cosmetics, b) changing dietary habits, c) getting patch test site wet, d) removing the patch, e) wearing tight or restrictive clothing that can remove patch, and f) engaging in activities that result in excessive sweating.
* A participant with current or recent (within last 6 months before the start of the study) history of atopic lesions and/or eczema.
* A participant with a history of allergic reactions to topical-use products, cosmetics or medications or their ingredients.
* A participant with any history of significant diseases or medical conditions known to alter skin appearance or physiologic response (e.g. uncontrolled diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* A participant considered immune-compromised.
* A participant with active dermatosis (local or disseminated) that might interfere with the results of the study.
* A participant currently using any medication which in the opinion of the investigator, may affect the evaluation of the investigational product or place the participant at undue risk.
* A participant who has used any of the following topical or systemic medications up to two weeks before the screening visit: immuno-suppressants, antihistamines, non-steroidal anti-inflammatory drugs (NSAIDS, high dose aspirin), and/or corticosteroids.
* A participant who has used a transcutaneous electrical nerve stimulation (TENS) machine 1 day before the screening visit.
* A participant who has used oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* A participant who has been vaccinated up to 1 month before the screening visit or is intending to receive a vaccination during their participation in the study.
* A participant with any skin marks on the back that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, open sores, pimples, cysts, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* A participant that intends bathing (in the sea or a pool), using sauna, or partaking in water sports, or activities that lead to intense sweating.
* A participant that is a prisoner or involuntary incarcerated.
* A participant from an indigenous tribe.
* A participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Brazil.
Pre-assignment Details: A total of 369 participants were screened, of which 302 participants were enrolled and 280 participants were randomized in induction phase and 258 participants went into the challenge phase.
Groups:
- Overall Participants: Participants applied a semi-occlusive adhesive patch containing the test products 0.02 milliliters per centimeters square (mL/cm^2) and 0.9% NaCl as negative control in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 minutes (min), test sites were evaluated as per the International Contact Dermatitis Research Group (ICDRG) scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
Period: Induction Phase
Arm/Group | Overall Participants
Started | 280
Completed | 258
Not Completed | 22
Not completed — (missed study visits) | 16
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 2
Period: Rest Phase
Arm/Group | Overall Participants
Started | 258
Completed | 258
Not Completed | 0
Period: Challenge Phase
Arm/Group | Overall Participants
Started | 258
Completed | 255
Not Completed | 3
Not completed — missed study visits | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of any study product.
Groups:
- Overall Participants: Participants applied a semi-occlusive adhesive patch containing the test products 0.02 mL/cm^2 and 0.9% NaCl as negative control in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 min, test sites were evaluated as per the ICDRG scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
Arm/Group | Overall Participants
Number analyzed (Participants) | 280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 241
  More than one race | 1
  Unknown or Not Reported | 0
Fitzpatrick Skin Type Grading [Number; unit: Number of Participants] — Fitzpatrick scale was used to classify participant's skin type by their response to sun exposure and confirm that participants were free of any pre-existing dermatological pathology.This scale emphasizes on potentials for irritation, burns and hyperpigmentation, indicators for future product choices. Scoring was done on scale I to VI, where I-always burns easily;never tans,II-always burns easily;tans minimally,III-burns moderately;tans gradually,IV-burns minimally, always tans well, V-rarely burns, tans profusely and VI-never burns. Higher score represents better results.
  Number of Participants
    I - Always burns easily, never tans (pale white skin) | 6
    II - Always burns easily; tans minimally (white skin) | 53
    III - Burns moderately; tans gradually (light brown skin) | 137
    IV - Burns minimally, always tans well (moderate brown skin) | 84
    V - Dark brown skin | 0
    VI - Deeply pigmented dark brown to black skin | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Potential Sensitisation Reactions as Assessed by Dermatologist on Day 40
Description: Human repeated insult patch test (HRIPT) reactions as per (ICDRG) were scored by trained blind evualuator on the scale of '- to +++', where '-':negative reaction,'?+':doubtful reaction; faint erythema only,'+': weak (non-vesicular) positive reaction;erythema, infiltration and possibly papules,'++': strong (vesicular) positive reaction; erythema, infiltration, papules and vesicles,'+++': extreme positive reaction; bullous reaction, intense erythema and infiltration, coalescing vesicles. Score '-' indicated no adverse reaction, whereas, '+++' indicated very strong adverse reaction. Any positive reaction (a score of '+' or greater) was considered as potential sensitization based upon dermatologist discretion. The assessment of positive reactions was determined by the blinded dermatologist and reported as Yes/ No/ Unable to determine. Percentage of participants with potential sensitization (count of "Yes"/ total reactions) were reported in form of numbers in this outcome measure.
Time Frame: Day 40
Population: The Safety Population comprised all randomized participants who received application of any of the study products.Number analyzed in this outcome measure signifies those who were evaluated.
Measure: Number; unit: Number of participants
Groups:
- Developmental Serum: Participants applied a semi-occlusive adhesive patch containing the developmental serum 0.02 mL/cm^2 in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 min, test sites were evaluated as per the ICDRG scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
- Developmental Lotion: Participants applied a semi-occlusive adhesive patch containing the developmental lotion 0.02 mL/cm^2 in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 min, test sites were evaluated as per the ICDRG scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
- Developmental Cream: Participants applied a semi-occlusive adhesive patch containing the developmental cream 0.02 mL/cm^2 in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 min, test sites were evaluated as per the ICDRG scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
- Negative Control: Participants applied a semi-occlusive adhesive patch containing 0.9% NaCl as negative control in an individual cell of the patch topically to the dorsum, repeatedly for 3 weeks (9 times) in induction phase (48 (+/-4) hours in weekdays and 72 (+/-4) hours in weekends. Patch was removed and area was gently wiped. After 30 min, test sites were evaluated as per the ICDRG scale. After 2 weeks of rest phase, participants followed the similar procedure with single application for 48 (+/-4) hours in the challenge phase. After 30 min, test sites were evaluated.
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 280 | 280 | 280 | 280
Number of participants | 2 | 1 | 1 | 0

2. Secondary Outcome: Percentage of Participants With a Positive Reaction Score (Score of '+' or Greater) as Assessed by a Trained Evaluator
Description: HRIPT reactions as per ICDRG were scored by trained blind evaluator on the scale of '- to +++', where '-':negative reaction,'?+':doubtful reaction; faint erythema only,'+': weak (non-vesicular) positive reaction;erythema, infiltration and possibly papules,'++': strong (vesicular) positive reaction; erythema, infiltration, papules and vesicles,'+++': extreme positive reaction; bullous reaction, intense erythema and infiltration, coalescing vesicles. Score '-' indicated no adverse reaction, whereas, '+++' indicated very strong adverse reaction. Any positive reaction (a score of '+' or greater) was considered as potential sensitization based upon dermatologist discretion. The assessment was determined by the blinded dermatologist and reported as a score of '+' or greater. Percentage of participants with any positive reaction (a score of '+' or greater) will be reported in numbers in this outcome measure.
Time Frame: Day 40
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 280 | 280 | 280 | 280
Number of participants
  Induction Phase | 4 | 4 | 4 | 4
  Challenge Phase: number analyzed (Participants) | 257 | 257 | 257 | 257
  Challenge Phase | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Upto Day 40
Description: The Safety Population included all randomized participants who received at least 1 dose of any study product. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported.
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/280 | 0/280 | 0/280 | 0/280 | 0/280
Serious Adverse Events (participants affected / at risk) | 1/280 | 1/280 | 1/280 | 1/280 | 1/280
Other Adverse Events (participants affected / at risk) | 12/280 | 12/280 | 12/280 | 12/280 | 12/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Developmental Serum (N=280) | Developmental Lotion (N=280) | Developmental Cream (N=280) | Negative Control (N=280) | Overall Participants (N=280)
Alcohol Poisoining (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Developmental Serum (N=280) | Developmental Lotion (N=280) | Developmental Cream (N=280) | Negative Control (N=280) | Overall Participants (N=280)
Headache (Nervous system disorders) | 4 (5) | 4 (5) | 4 (5) | 4 (5) | 4 (5)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT04007159/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04007159/SAP_001.pdf